CLINICAL TRIAL: NCT00393848
Title: Restoration of Muscle Following Hip Surgery
Brief Title: Effectiveness of Two Types of Treatment in Restoring Muscle After Hip or Knee Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01AR052293 (NIH); 70451; 1R01AR052293-01A2 (NIH)
Record Dates: First submitted 2006-10-27; First posted 2006-10-30 (Estimated); Results first posted 2014-06-02 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2014-05

CONDITIONS: Hip Fracture; Osteoarthritis; Femur Head Necrosis
Keywords: Hip Replacement Arthroplasty; Hip Replacement Surgery; Hip Surgery; Hip Rehabilitation; Avascular Necrosis; Knee replacement surgery; Total knee arthroplasty
MeSH Terms: conditions — Hip Fractures; Osteoarthritis; Femur Head Necrosis; Osteonecrosis | interventions — Ketoconazole

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Experiment 2 - Experimental Group (Experimental)
  Interventions: Drug: Ketoconazole
- Experiment 1 - Standard of care Group (No Intervention)
- Experiment 1 - Experimental Group (Experimental)
  Interventions: Drug: Essential amino acid supplement
- Experiment 2 - Placebo Group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Essential amino acid supplement — 15g of essential amino acid in capsule form three times daily during hospitalization, continued through 6 weeks after discharge.
  Arms: Experiment 1 - Experimental Group
Drug: Ketoconazole — 200mg ketoconazole twice daily; started night before surgery and continued through hospitalization.
  Arms: Experiment 2 - Experimental Group
Drug: Placebo — Placebo for Ketoconazole
  Arms: Experiment 2 - Placebo Group

SUMMARY:
The purpose of this study is to determine the effects of two postoperative interventions designed to preserve muscle protein after major hip or knee surgery.

DETAILED DESCRIPTION:
Hip fractures among the elderly are a major health concern. Nearly one-third of elderly hip fracture patients die within 1 year of the injury. Events surrounding the actual injury and any necessary surgical repair often lead to reduced muscle protein, and eventually, muscle strength. Loss in everyday function and independence may follow, especially in elderly or frail individuals. The decrease in protein synthesis may be caused by two main events following injury and surgery: prolonged inactivity and an increase in stress hormone levels. Preventing a loss in protein may help to improve outcomes for individuals undergoing hip surgery and rehabilitation. The purpose of this study is to determine the effects of two postoperative interventions designed to retain muscle protein after major hip or knee surgery in adults.

This study will include two experiments. Experiment 1 will include individuals who are scheduled for hip or knee replacement surgery because of osteoarthritis (the need to repair or replace the affected joint), or avascular necrosis (bone tissue death caused by lack of blood supply). Experiment 1 participants will be randomly assigned to one of two groups:

* Group 1 participants will receive daily supplements of essential amino acids, which are thought to stimulate protein synthesis.
* Group 2 participants will receive standard rehabilitation care while in the hospital and will serve as controls for the effect of time on recovery.

Participants will be in the hospital for about 4 days. On the morning of surgery, blood and urine collection will occur. During surgery, substances called tracers, measuring the extent of protein synthesis and breakdown, will be injected into a vein for the first metabolic study. Additional blood and muscle samples will also be taken. After surgery, when participants arrive in the surgical recovery unit and are able to eat, they will begin to record all food intake and will receive their assigned treatment. Treatment, in the form of gel capsules, will be taken 2.5 hours after each meal. Urine will be collected throughout hospitalization and blood will be collected each morning. Prior to discharge, a 24-hour metabolic study will be performed, including tracer injections and muscle biopsies. After discharge, participants will be provided with 6 weeks' worth of their assigned treatment. Follow-up visits will occur 2 and ~6 to 8 weeks after surgery. These visits will include various muscle function and physical performance tests. Participants will also undergo a dual energy x-ray absorptiometry (DEXA) scan, which will be used to determine muscle mass.

Experiment 2 participants will include individuals scheduled for either hip or knee replacement surgery or fracture repair surgery. Participants will be randomly assigned to one of two groups:

* Group 1 participants will receive the antifungal drug ketoconazole, which is thought to reduce levels of the stress hormone cortisol.
* Group 2 participants will receive placebo and standard rehabilitation care while in the hospital.

Participants will begin taking their assigned treatments the day prior to surgery; those with a hip fracture will take their assigned treatment at least 4 hours prior to surgery. The same procedures that occurred in Experiment 1 during surgery and hospitalization will be carried out during Experiment 2. The second metabolic study, however, will last only 1 hour and will include a standard clinical meal.

ELIGIBILITY:
Inclusion Criteria for All Participants:

* Scheduled for surgery because of osteoarthritis, avascular necrosis, fracture, or revision of total joint replacement in the hip or knee

Exclusion Criteria for All Participants:

* Taking insulin, thiazolidinediones (TZD), or metformin
* Kidney insufficiency, as indicated by serum creatinine of more than 2.0 mg/dl
* Recently treated cancer other than basal cell carcinoma
* Any other condition or event that would be considered as reason for exclusion by the study investigators
* Pregnancy

Exclusion Criteria for Experiment 1 Participants:

* Severe hypertension as indicated by requiring more than two drugs for blood pressure control
* History of hypo- or hypercoagulation disorders, including individuals who have taken warfarin (Coumadin)
* Atrial fibrillation, angina, or congestive heart failure

Exclusion Criteria for Experiment 2 Participants:

* Liver disease or abnormal liver function tests
* HIV infected
* Active hepatitis
* Any uncontrolled metabolic disease, including liver or kidney disease
* Taking medications that use the cytochrome P450 pathway for metabolism and unable to discontinue their use for the duration of the study
* Require certain medications. More information on this criterion can be found in the protocol.
* Gastrointestinal absorption disorders that affect nutrient uptake

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arny Ferrando, PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Experiment 1 - Amino Acid Supplement: Essential amino acid supplement : 15g of essential amino acid in capsule form three times daily during hospitalization, continued through 6 weeks after discharge.
- Experiment 1 - Standard of Care: Usual clinical care with no dietary intervention.
- Experiment 2 - Ketoconazole: 200mg ketoconazole twice daily; started night before surgery and continued through hospitalization.
- Experiment 2 - Placebo: Placebo for Ketoconazole twice daily; started night before surgery and continued through hospitalization.
Period: Overall Study
Arm/Group | Experiment 1 - Amino Acid Supplement | Experiment 1 - Standard of Care | Experiment 2 - Ketoconazole | Experiment 2 - Placebo
Started | 16 | 9 | 6 | 9
Completed | 16 | 9 | 4 | 8
Not Completed | 0 | 0 | 2 | 1
Not completed — Surgical schedule | 0 | 0 | 0 | 1
Not completed — Personal reasons | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Experiment 1 - Standard of Care: Usual clinical care - no dietary intervention.
- Total: Total of all reporting groups
Arm/Group | Experiment 1 - Amino Acid Supplement | Experiment 1 - Standard of Care | Experiment 2 - Ketoconazole | Experiment 2 - Placebo | Total
Number analyzed (Participants) | 16 | 9 | 4 | 8 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 7 | 4 | 7 | 31
  >=65 years | 3 | 2 | 0 | 1 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (7) | 56 (8) | 44 (15) | 46 (15) | 51 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 2 | 2 | 14
  Male | 9 | 6 | 2 | 6 | 23
Region of Enrollment [Number; unit: participants]
  United States | 16 | 9 | 4 | 8 | 37

OUTCOME MEASURES:

1. Primary Outcome: Muscle Protein Synthesis
Time Frame: Perioperative and discharge
Measure: Mean (Standard Error); unit: %/d
Groups:
- Experiment 1 - Standard of Care: Usual clinical care without dietary intervention
Arm/Group | Experiment 1 - Amino Acid Supplement | Experiment 1 - Standard of Care | Experiment 2 - Ketoconazole | Experiment 2 - Placebo
Number analyzed (Participants) | 16 | 9 | 4 | 8
%/d
  Perioperative MPS | 1.38 (0.12) | 0.84 (0.11) | 1.42 (0.48) | 1.36 (0.22)
  Discharge MPS | 1.23 (0.16) | 1.49 (0.18) | NA (NA) — Not performed | NA (NA) — Not performed

2. Secondary Outcome: Change in Maximal Voluntary Contraction
Time Frame: Baseline and 6 weeks post surgery
Population: Measure not performed in Experiment 2
Measure: Mean (Standard Error); unit: kg/kg leg lean mass
Arm/Group | Experiment 1 - Amino Acid Supplement | Experiment 1 - Standard of Care
Number analyzed (Participants) | 16 | 9
kg/kg leg lean mass | 0.68 (0.3) | 0.34 (0.32)

ADVERSE EVENTS:
Groups:
- Experiment 1 - Amino Acid Supplement: Essential amino acid supplement: 15g of essential amino acid in capsule form three times daily during hospitalization, continued through 6 weeks after discharge.
Arm/Group | Experiment 1 - Amino Acid Supplement | Experiment 1 - Standard of Care | Experiment 2 - Ketoconazole | Experiment 2 - Placebo
Serious Adverse Events (participants affected / at risk) | 0/16 | 1/9 | 0/6 | 0/9
Other Adverse Events (participants affected / at risk) | 0/16 | 0/9 | 0/6 | 0/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experiment 1 - Amino Acid Supplement (N=16) | Experiment 1 - Standard of Care (N=9) | Experiment 2 - Ketoconazole (N=6) | Experiment 2 - Placebo (N=9)
Mastectomy for breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No